CLINICAL TRIAL: NCT06517004
Title: An Open-label, Single-arm Study of JWCAR201 in the Treatment of Relapsed or Refractory Diffuse Large B-cell Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Rong Tao, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JWCAR201002
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: CAR-T therapy; Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JWCAR201 Treatment Arm (Experimental): Patients will be administrated with autologous CD19/CD20-directed CAR-T cells after lymphocyte depletion by fludarabine and cyclophosphamide.
  Interventions: Biological: JWCAR201

INTERVENTIONS:
Biological: JWCAR201 — Autologous CD19/CD20-directed CAR-T cells, single infusion intravenously

SUMMARY:
This is an open-label, single-arm study to investigate the efficacy and safety signals of JWCAR201 amongst subjects with relapsed or refractory diffuse large B-cell lymphoma (DLBCL).

DETAILED DESCRIPTION:
This is an open-label, single-arm, investigator-initiated study (IIT) to evaluate the safety an JWCAR201 in adult patients with relapsed/refractory diffuse large B-cell lymphoma (r/r DLBCL). The study employs a two-stage, Continual Reassessment Method (CRM)-like dose escalation design. In the first stage, each dose cohort will use an accelerated titration approach, escalating to the dose level at which a Dose-Limiting Toxicity (DLT) occurs or the 50 × 10^6 CAR+ T-cell dose level (whichever is reached first). The second stage will start at observed DLT dose level or the 50^6 CAR+ T-cell dose level, an model-based CRM method using a single-parameter Logistic model will be used to describe the relationship between the JWCAR201 dose and the probability of observed DLTs. The Maximum Tolerated Dose (MTD) is defined as the highest an estimated DLT probability below the 25% target toxicity level. For each dose level, a prior mean DLT risk (skeleton) will be set based on historical data. After enrolling ≥3 patients perort, the prior DLT risk will be updated based on the available study data, and the DLT risk will be communicated to the Data Safety Monitoring Committee to recommend the next cohort dose. The study plans to start at 25 × 10^6 CAR+ T cells as the initial dose, with exploration across three dose levels (25 × 10^6, 50 × 10^6, 75 × 10^6 CAR+ T cells), and 15 × 10^6 CAR+ T cells or lower and 100 × 10^6 CAR+ T cells or higher as backup doses, aiming to evaluate the safety, tolerability of JWCAR201 in r/r DLBCL and determine the recommended dose for expansion. Additionally, pharmacokinetic and pharmacodynamic characteristics are also study objectives.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18
2. Voluntarily willing to participate in the study and sign the written informed consent form
3. Histologically confirmed diffuse large B-cell lymphoma (DLBCL) with immunohistochemistry (IHC) CD20-positive
4. Patients must be priorly treated by Anthracyclines and anti-CD20-targeted regimens, and must be refractory or relapsed to at least ≥2 treatment lines of standard of care or autologous hematopoietic stem-cell transplantation (HSCT)
5. At least one measurable lesion by CT or PET per Lugano criteria
6. Eastern Cooperative Oncology Group (ECOG) performance status scale ≤1
7. Adequate organ functions
8. Adequate venous access for apheresis
9. Women of childbearing potential must agree to use an effective and reliable contraceptive method till 1-year post-infusion
10. Male patients who have not undergone vasectomy and have sexual activity with women of childbearing potential must agree to the use of a barrier contraceptive till 1-year post-infusion

Exclusion Criteria:

1. Primary central nervous system lymphoma
2. Another primary malignancy within 2 years
3. Active infections of hepatitis B virus (HBV), hepatitis C virus (HCV), human immunodeficiency virus (HIV), or syphilis
4. With severe active deep venous thrombosis or pulmonary embolism within 3 months
5. Treated with anti-coagulations (except for prophylaxis use) due to severe active deep venous thrombosis or pulmonary embolism within 3 months
6. Uncontrolled or active infection
7. Acute or chronic graft-versus-host disease (GvHD)
8. With severe cardiovascular diseases within 6 months
9. With severe clinically-significant central nervous system disorders within 6 months
10. Pregnant or lactating women
11. Not satisfying pre-defined wash-out period for apheresis
12. Unable or unwilling to comply with the study protocol, judged by the investigator, or other situations implying that the subject might not be appropriate to participate in the study
13. Previously treated with any genetically engineered modified T-cell therapy nor other cell-gene therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2024-07-18 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Rate of dose-limiting toxicities (DLTs) | 28 days
  Dose limiting toxicities for each subject
AE/SAE | 24 months
  Incidence and severity of adverse events (AE), and serious adverse event (SAE)

SECONDARY OUTCOMES:
Copy number of the vector transgene of JWCAR201 in peripheral blood | 24 months
  The pharmacokinetic parameters of JWCAR201 will be evaluated by quantitative polymerase chain reaction (qPCR) for the copy number of the vector transgene of JWCAR201 in peripheral blood to evaluate T-cell expansion and persistence.
CD19-positive cells and CD20-positive cells in peripheral blood | 24 months
  CD19-positive cells and CD20-positive cells in peripheral blood will be tested by flow cytometry (FCM).
Objective response rate (ORR) | 24 months
  Proportion of patients whose tumor volume has reached a predetermined value and can maintain a minimum time limit, including complete response and partial response patients.
Complete response rate (CRR) | 24 months
  The percentage of patients with advanced or metastatic cancer who have achieved complete response to a therapeutic intervention in clinical trials of anticancer agents.
Duration of response (DOR) | 24 months
  The time from the date of first response (PR or better) to the date of disease progression or death after JWCAR201 infusion.
Progression-free survival (PFS) | 24 months
  The time from JWCAR201 infusion to the date of progression as assessed by Lugano criteria or death.
Overall survival (OS) | 24 months
  Defined as the time from the date of first infusion of JWCAR201 to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Rong Tao, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No